CLINICAL TRIAL: NCT07258186
Title: Feasibility Study of the Generation of Endometrial Carcinoma Organoids From Tumor Samples Transferred From Extramural Facilities
Brief Title: Generation of Endometrial Carcinoma Organoids
Acronym: organoids endo
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: RS316/IRE/25
Record Dates: First submitted 2025-11-18; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tumor and peri-tumor tissues
  Blood (Serum and PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with endometrial cancer of the endometrioid histology at any stage of the disease.: Patients aged 18 years and older with a histological diagnosis of endometrial cancer of the endometrioid histology at any stage of disease (FIGO I-IV), recurrence/metastasis from endometrial endometrioid cancer, who are candidates for surgery or hysterectomy and who will undergo surgery after signing an informed consent form, will be prospectively recruited.
  Interventions: Genetic: Generation of organoids from endometrial tumor tissue collected during surgery, performed according to standard clinical practice

INTERVENTIONS:
Genetic: Generation of organoids from endometrial tumor tissue collected during surgery, performed according to standard clinical practice — Creation of endometrial carcinoma organoids from tumor tissue from extramural structures, verifying the feasibility of organoid generation. Evaluate the impact of sample transport and storage conditions on the success of the process, considering the challenges associated with preserving tissue integrity.

SUMMARY:
A prospective pilot genetic study to evaluate the feasibility of generating organoids from endometrial tumor tissue collected during surgery, performed according to standard clinical practice. Samples will be collected from collaborating extramural facilities, with the aim of analyzing the impact of transport on tissue viability and the success of organoid culture. This study is for exploratory purposes only, without altering the diagnostic and therapeutic pathways of the participants.

DETAILED DESCRIPTION:
The prospective study involves the collection and freezing of biological samples at the IRE Translational Oncology Research Unit. Collecting and using:

* Fresh tissue: tumor and peritumor tissue from the same patient, obtained surgically at participating centers, will be collected under the supervision of a dedicated pathologist, sent to the IRE Translational Oncology Research Unit, and frozen. The collected tissue will be processed and used to perform gene expression profiling using RNAseq and WES and to generate organoids.
* Blood (Serum and PBMCs) - A blood sample (EmoT0) will also be collected for each patient before surgery. This sample will be used to prepare serum for aliquoting/freezing, and peripheral blood mononuclear cells (PBMCs). These will also be sent, frozen, and stored at the IRE Translational Oncology Research Unit. These will be used to evaluate the organoids' response to immunotherapy treatments through coculture experiments.

Only biological material whose availability and suitability are guaranteed will be used to archive appropriate material as required by law. It will then be sent to the research laboratories of the IRE Translational Oncology Research Unit and will be used for genomic analysis and the generation of organoids.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Patients with a histological diagnosis of: endometrial cancer, endometrioid histology, any stage of disease (FIGO I-IV), recurrence/metastasis from endometrial endometrioid cancer, and candidates for surgery and/or hysterectomy;
* Written informed consent (study participation and data processing) must be obtained in person and/or through a legal representative/guardian/support administrator/witness, before any study-specific procedure is performed.

Exclusion Criteria:

* Comorbidities not controlled with adequate medical therapy;
* Endometrial cavity infections (pyometra);
* Synchronous tumors;
* Neoadjuvant treatments;
* Previous radiation treatments to the pelvic region.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Patients with a histological diagnosis of endometrioid endometrial cancer at any stage of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-23 (Actual); Primary Completion 2028-09-23 (Estimated); Study Completion 2028-09-23 (Estimated)

PRIMARY OUTCOMES:
Feasibility of organoid generation | 42 months
  The feasibility of generating endometrial carcinoma organoids from tumor tissue will be assessed by analyzing the success rate in organoid generation, expressed as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS National Cancer Institute "Regina Elena", Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided